CLINICAL TRIAL: NCT01842009
Title: Single-arm, Open-label, Phase II Trial of HD-tDCS in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: ElMindA Ltd (Industry)
Responsible Party: Principal Investigator, Felipe Fregni, Associate Professor, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013P000384
Record Dates: First submitted 2013-04-18; First posted 2013-04-29 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Fibromyalgia; Chronic Pain
Keywords: transcranial stimulation; direct current
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Active anodal HD-tDCS (Experimental): Subjects will undergo 20 minutes active HD-tDCS.
  Interventions: Device: High Definition transcranial Direct Current Stimulation

INTERVENTIONS:
Device: High Definition transcranial Direct Current Stimulation
  Other Names: 4X1 low-intensity direct current stimulator

SUMMARY:
The purpose of this study is to investigate the mean number of stimulation (high definition-transcranial direct current stimulation) sessions (up to 26) needed to achieve a clinical response with this response defined as a 50% decrease in Visual Analog Scale (VAS) for pain. These data will be important in defining the optimal number of sessions for future fibromyalgia subjects in Phase III trials.

ELIGIBILITY:
Inclusion Criteria:

* Providing informed consent to participate in the study
* 18 to 85 years old, both male and female
* Have a diagnosis of Fibromyalgia
* Existing pain for more than 3 months with an average of at least 4 on a 0-10 VAS scale
* Pain resistant to common analgesics and medications for chronic pain such as Tylenol, Aspirin, Ibuprofen, Soma, Parafon Forte DCS, Zanaflex and Codeine.

Exclusion Criteria:

* Pregnancy
* Contraindications to tDCS: metal in the head or implanted brain medical devices
* History of alcohol or drug abuse within the past 6 months as self-reported
* Use of carbamazepine within the past 6 months as self-reported
* Severe depression (with a score of >30 in the Beck Depression Inventory)
* Any history of epilepsy, stroke, moderate-to-severe traumatic brain injury or severe migraines
* History of unexplained fainting spells as self-reported
* Neurosurgery as self-reported

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2016-06-07 (Actual)

PRIMARY OUTCOMES:
Mean number of sessions needed to achieve 50% decrease in Visual Analogue Scale (VAS) | approximately 4.5 months
  Investigate the mean number of sessions (up to 26) needed to achieve clinical response associated with the use of HD-tDCS over the primary motor cortex (M1), with response defined at a 50% decrease in baseline Visual Analogue Scale (VAS) for pain.

SECONDARY OUTCOMES:
Number of subjects who achieve clinical response | Approximately 4.5 months
  We will count the number of subjects who achieve clinical response (as defined in Aim 1 as a 50% reduction in baseline VAS) for the duration of the trial.
Measurement of sensory and auditory evoked potentials | Approximately 4.5 months
  We will measure brain pain response using electroencephalography (EEG) to measure somatosensory Event Related Potentials (ERPs) with a heat pain threshold device. We will also measure auditory ERPs. We will investigate the relationship between these ERP measurements and overall clinical response of patients (as outlined in Aim 1 and Aim 2)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD PhD MPH, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Charlestown, Massachusetts, United States

REFERENCES:
- [Derived] Castillo-Saavedra L, Gebodh N, Bikson M, Diaz-Cruz C, Brandao R, Coutinho L, Truong D, Datta A, Shani-Hershkovich R, Weiss M, Laufer I, Reches A, Peremen Z, Geva A, Parra LC, Fregni F. Clinically Effective Treatment of Fibromyalgia Pain With High-Definition Transcranial Direct Current Stimulation: Phase II Open-Label Dose Optimization. J Pain. 2016 Jan;17(1):14-26. doi: 10.1016/j.jpain.2015.09.009. Epub 2015 Oct 9. PMID 26456677